CLINICAL TRIAL: NCT00006114
Title: First Line Treatment of Metastatic Hormone Refractory Prostate Cancer With a Combination of Novantrone-Navelbine
Brief Title: Combination Chemotherapy in Treating Patients With Metastatic Prostate Cancer That Has Not Responded to Hormone Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068126; FRE-GERCOR-NONA-U98-1; EU-20025
Record Dates: First submitted 2000-08-03; First posted 2003-01-27 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2000-09

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Mitoxantrone; Vinorelbine

INTERVENTIONS:
Drug: mitoxantrone hydrochloride
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients who have metastatic prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of the combination of mitoxantrone and vinorelbine in terms of response rate, progression free survival, overall survival, and quality of life in patients with metastatic hormone refractory adenocarcinoma of the prostate.
* Determine the toxicities of this treatment regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive vinorelbine IV on days 1 and 8 and mitoxantrone IV on day 8. Treatment repeats every 3 weeks for up to 9 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed prior to treatment, prior to each course, and then at 2 months after study completion.

Patients are followed every 3 months until disease progression.

PROJECTED ACCRUAL: A total of 14-39 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed stage IV hormone refractory adenocarcinoma of the prostate
* Progressive disease despite hormonal therapy or orchiectomy
* No brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 to 80

Performance status:

* WHO 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Absolute neutrophil count at least 2,000/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 9 g/dL

Hepatic:

* Alkaline phosphatase no greater than 2 times upper limit of normal (ULN) (unless bone metastasis)
* Bilirubin less than 2 times ULN

Renal:

* Creatinine less than 2 times ULN

Cardiovascular:

* Adequate cardiac function

Other:

* No other prior malignancy except curatively treated basal or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* See Disease Characteristics
* Prior corticosteroids allowed if started at least 8 weeks prior to study

Radiotherapy:

* At least 8 weeks since prior extensive radiotherapy

Surgery:

* See Disease Characteristics

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-05

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Wendling, MD, Study Chair — Centre Hospitalier Intercommunal Toulon - La Seyne Sur Mer
Locations (10):
- France (10):
  - Hopital Saint-Louis, Amiens
  - Hopital Gouin, Clichy
  - Hopital Perpetuel Secours, Levallois-Perret
  - CHU de la Timone, Marseille
  - Hopital Laennec, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Tenon, Paris
  - Polyclinique De Courlancy, Reims
  - C.H. Senlis, Senlis
  - Centre Hospitalier Intercommunal Toulon - La Seyne/Mer, Toulon